CLINICAL TRIAL: NCT04185090
Title: An Open-label, Single or Multiple-dose, Fixed-sequence, 3-treatment, 3-Period Phase 1 Study to Evaluate the Pharmacokinetic/Pharmacodynamic Interactions and Safety Between ID1801 and ID1803 in Healthy Male Subjects
Brief Title: To Evaluate the Pharmacokinetic/Pharmacodynamic Interactions and Safety Between ID1801 and ID1803 in Healthy Male Adults
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ID-VARE-101
Record Dates: First submitted 2019-11-28; First posted 2019-12-04 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-11

CONDITIONS: Hypertension; Dyslipidemias
MeSH Terms: conditions — Hypertension; Dyslipidemias

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ID1801 (Active Comparator): qd daily for 6days Intervention: Drug: administration of ID1801 for 6days.
  Interventions: Combination Product: ID1801
- ID1803 (Active Comparator): qd daily for 10days Intervention: Drug: administration of ID1803 for 10days.
  Interventions: Combination Product: ID1803
- ID1801 and ID1803 (Experimental): qd daily for 7days Intervention: Drug: administration of ID1801 and ID1803.
  Interventions: Combination Product: ID1803+ID1801

INTERVENTIONS:
Combination Product: ID1803 — Amlodipine 10mg/Valsartan 160mg
  Arms: ID1803
Combination Product: ID1801 — Ezetimibe 10mg/Rosuvastatin Ca 20.8mg
  Arms: ID1801
Combination Product: ID1803+ID1801 — Amlodipine 10mg/Valsartan 160mg Ezetimibe 10mg/Rosuvastatin Ca 20.8mg
  Arms: ID1801 and ID1803

SUMMARY:
This study is designated to evaluate the pharmacokinetic interactions of valsartan, amlodipine besylate, rosuvastatin, and ezetimibe in healthy male volunteers.

DETAILED DESCRIPTION:
An Open-label, Single or Multiple-dose, Fixed-sequence, 3-treatment, 3-Period phase 1 study to Evaluate the Pharmacokinetic/Pharmacodynamic Interactions and Safety between ID1801 and ID1803 in Healthy Male Subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male volunteers aged 19 to 45 years
* Subjects who have over 50kg and BMI more than 18.5kg/m2 and less than 29.9kg/m2
* Males must be agree to practice a medically acceptable method* of birth control and will not donate sperm during the study.
* Subjects who provided written informed consent to participate in this study and voluntarily taken part in during the entire study period

Exclusion Criteria:

* Subject with serious active cardiovascular, respiratory, hepatologic, renal, hematologic, gastrointestinal, immunologic, dermal, neurologic, or psychological disease or history of such disease
* Subject with symptoms of acute disease within 28days prior to study medication dosing
* Medical history or evidence that can affect absorption, distribution, metabolism and excretion of a given drug
* Drugs or other drugs (aspirin, antibiotics, etc.) that contain the following drug categories or components of the same strain have an overactive or clinically significant history of hypersensitivity:
* Subject with a history of drug abuse or urinalysis positive
* Subject with clinically significant active chronic disease
* Subject with genetic problems such as galactose intolerance, Lapp lactose deficiency or glucose-galactose malabsorption.
* Genetic myopathic disorder or related family history
* Positive test results for HBs Ab, HCV Ab, Anti HIV(AIDS), RPR Ab
* Subject with clinically significant allergic disease (except for mild allergic rhinitis and mild allergic dermatitis that are not needed to administer drug)
* Subject who cannot take standard meal in hospitalization
* Present history of hypothyroidism or clinically significant assay
* Subjects who donated whole blood or partial blood within 2 or 1 month, respectively, prior to the first administration.
* Subject taking inducer or inhibitor of drug metabolism enzyme such as barbital within 30days prior to study medication dosing
* Smokers whose average daily smoking amount exceeds 10 cigarettes per day within 3 months before the first dosing day and those who can't quit from 48 hours before dosing to the time of the last blood sampling.
* Subjects who judged ineligible by the investigator

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-02 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
AUCτ(Amlodipine, valsartan, rosuvastatin, free ezetimibe) | 0~72hours
  Amlodipine, valsartan, rosuvastatin, free ezetimibe: AUCτ
Cmax,ss(Amlodipine, valsartan, rosuvastatin, free ezetimibe) | 0~72hours
  Amlodipine, valsartan, rosuvastatin, free ezetimibe: Cmax,ss

SECONDARY OUTCOMES:
AUCτ(N-desmethyl rosuvastatin, total ezetimibe) desmethyl rosuvastatin, total ezetimibe: AUCτ, Cmax,ss | 0~72hours
  N-desmethyl rosuvastatin, total ezetimibe: AUCτ
Cmax,ss(N-desmethyl rosuvastatin, total ezetimibe) desmethyl rosuvastatin, total ezetimibe: AUCτ, Cmax,ss | 0~72hours
  N-desmethyl rosuvastatin, total ezetimibe: Cmax,ss
Cmin,ss(amlodipine, valsartan, rosuvastatin, N-desmethyl rosuvastatin, free ezetimibe and, total ezetimibe) | 0~72hours
  amlodipine, valsartan, rosuvastatin, N-desmethyl rosuvastatin, free ezetimibe and, total ezetimibe: Cmin,ss
Tmax,ss(amlodipine, valsartan, rosuvastatin, N-desmethyl rosuvastatin, free ezetimibe and, total ezetimibe) | 0~72hours
  amlodipine, valsartan, rosuvastatin, N-desmethyl rosuvastatin, free ezetimibe and, total ezetimibe: Tmax,ss
t1/2(amlodipine, valsartan, rosuvastatin, N-desmethyl rosuvastatin, free ezetimibe and, total ezetimibe) | 0~72hours
  amlodipine, valsartan, rosuvastatin, N-desmethyl rosuvastatin, free ezetimibe and, total ezetimibe: t1/2
CLss/F(amlodipine, valsartan, rosuvastatin, N-desmethyl rosuvastatin, free ezetimibe and, total ezetimibe) | 0~72hours
  amlodipine, valsartan, rosuvastatin, N-desmethyl rosuvastatin, free ezetimibe and, total ezetimibe: CLss/F
Vd/F(amlodipine, valsartan, rosuvastatin, N-desmethyl rosuvastatin, free ezetimibe and, total ezetimibe) | 0~72hours
  amlodipine, valsartan, rosuvastatin, N-desmethyl rosuvastatin, free ezetimibe and, total ezetimibe: Vd/F
PTF(amlodipine, valsartan, rosuvastatin, N-desmethyl rosuvastatin, free ezetimibe and, total ezetimibe) | 0~72hours
  amlodipine, valsartan, rosuvastatin, N-desmethyl rosuvastatin, free ezetimibe and, total ezetimibe: PTF